CLINICAL TRIAL: NCT00868413
Title: A Phase 1 Study Evaluating the Safety of ABT-263 in Combination With Either Fludarabine/Cyclophosphamide/Rituximab (FCR) or Bendamustine/Rituximab (BR) in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Study of ABT-263 When Administered in Combination With Either Fludarabine/Cyclophosphamide/Rituximab or Bendamustine/Rituximab in Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-458
Record Dates: First submitted 2009-03-20; First posted 2009-03-25 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — navitoclax; fludarabine; Cyclophosphamide; Rituximab; Bendamustine Hydrochloride

ARMS (2):
- A (Active Comparator): FCR+ABT-263
  Interventions: Drug: ABT-263; Drug: FCR
- B (Active Comparator): BR+ABT-263
  Interventions: Drug: ABT-263; Drug: BR

INTERVENTIONS:
Drug: ABT-263 — ABT-263 is taken orally once daily for 3 days out of each 28 day cycle. This is a dose escalation study, therefore the dose of ABT-263 will change throughout the study.
Drug: FCR — Rituximab will be given by intravenous infusion for 1 day out of each 28 day cycle; Fludarabine will be given by intravenous infusion for 3 days out of each 28 day cycle; and Cyclophosphamide will be given by intravenous infusion for 3 days out of each 28 day cycle
  Other Names: fludarabine, cyclophosphamide, rituximab
  Arms: A
Drug: BR — Rituximab will be given by intravenous infusion for 2 days out of each 28 day cycle and Bendamustine will be given by intravenous infusion for 2 days out of each 28 day cycle
  Other Names: bendamustine, rituximab
  Arms: B

SUMMARY:
This is a Phase 1 study evaluating the safety of ABT-263 administered in combination with either FCR or BR in subjects with relapsed or refractory chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Must have relapsed or refractory Chronic Lymphocytic Leukemia (CLL), received no more than 5 prior myelosuppressive/chemotherapy regimens and must be a candidate for treatment with either Fludarabine/Cyclophosphamide/Rituximab (FCR) or Bendamustine/Rituximab (BR);
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of </=1;
* Must have adequate bone marrow independent of growth factor support (with the exception of subjects with bone marrow heavily infiltrated with underlying disease [80% or more] who may use growth factor support to achieve Absolute Neutrophil Count (ANC) eligibility criteria), per local laboratory reference range at Screening as follows: ANC >/=1000/mcL, Platelets>/= 100,000/mm3 (entry platelet count must be independent of transfusion within 14 days of Screening),Hemoglobin >/= 9.0 g/dL.

Exclusion Criteria:

* Subject has history or is clinically suspicious for cancer-related Central Nervous System disease;
* Has history of severe allergic or anaphylactic reactions to human, humanized, chimeric or murine monoclonal antibodies;
* Has undergone an allogeneic stem cell transplant; Exhibits evidence of other uncontrolled condition(s) including, but not limited to: uncontrolled systemic infection, diagnosis of fever and neutropenia within 1 week prior to study drug administration;
* Has underlying, predisposing condition of bleeding or currently exhibits signs of bleeding; Has a recent history of non-chemotherapy induced thrombocytopenic associated bleeding;
* Currently receiving or requires anticoagulation therapy;
* Has active immune thrombocytopenic purpura (ITP) or a history of being refractory to platelet transfusions (within 1 year prior to 1st dose of study drug);
* Has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile, characterize pharmacokinetics, and determine the MTD and recommended Phase 2 dose (RPTD) of ABT-263 when administered in combination with either FCR or BR in subjects with relapsed or refractory CLL. | Safety assessments = 1 wk, Pharmacokinetic (PK) Sampling = 1 wk for 1st 2 cycles, then, every other cycle starting Cycle 3 to Cycle 9, Determination of MTD & RPTD = Every 60 days

SECONDARY OUTCOMES:
Evaluate preliminary data regarding progression-free survival (PFS), tumor response rate and overall survival (OS) when ABT-263 is administered in combination with either FCR or BR. | Every 2 months
  Tumor assessments

CONTACTS AND LOCATIONS:
Overall Officials: Sari Enschede, MD, Study Director — AbbVie
Locations (6):
- United States (6):
  - Site Reference ID/Investigator# 17841, La Jolla, California
  - Site Reference ID/Investigator# 25899, Stanford, California
  - Site Reference ID/Investigator# 21622, Baltimore, Maryland
  - Site Reference ID/Investigator# 21621, Columbus, Ohio
  - Site Reference ID/Investigator# 39613, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 17943, Houston, Texas